CLINICAL TRIAL: NCT05980572
Title: Mobile Device Based Telerehabilitation for Frozen Shoulder-A Prospective Randomized Controlled Study.
Brief Title: Effects of App-assisted Home Exercise Program in Patients With Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chih-Chi ,Chen, Principle investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Defrozen_Shoulder_App
Record Dates: First submitted 2022-11-21; First posted 2023-08-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2022-08

CONDITIONS: Frozen Shoulder
Keywords: Frozen shoulder; App; Exercise
MeSH Terms: conditions — Bursitis; Alzheimer Disease; Motor Activity | interventions — Anti-Inflammatory Agents, Non-Steroidal; aceclofenac

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor blind to the arm of the subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- App intervention group (Experimental): Patients will receive instructions on performing the seven sets of frozen shoulder exercises mentioned earlier. The APP intervention group will be guided through the exercises using the mobile app. Each set of exercises will involve 10 repetitions, and it is recommended to perform four sessions per day.
  Interventions: Drug: Glenohumeral joint and subacromial space triamcinolone injections; Device: App-assisted exercise; Drug: Nonsteroidal anti-inflammatory drugs (aceclofenac)
- Conventional group (Active Comparator): patients will receive instructions on performing the seven sets of frozen shoulder exercises mentioned earlier. The conventional group will be provided with a printed pamphlet illustrating the exercises. Each set of exercises will involve 10 repetitions, and it is recommended to perform four sessions per day.
  Interventions: Drug: Glenohumeral joint and subacromial space triamcinolone injections; Drug: Nonsteroidal anti-inflammatory drugs (aceclofenac)

INTERVENTIONS:
Drug: Glenohumeral joint and subacromial space triamcinolone injections — All patients will receive both glenohumeral joint and subacromial space injections. The injections will consist of a solution containing 1 ml of 40 mg/ml triamcinolone acetonide and 1 ml of 1% lidocaine in each site. The glenohumeral joint injection will be performed blindly using an anterior approach. The needle will be inserted medially to the head of the humerus, located approximately 1 cm lateral to the coracoid process, and directed posteriorly at a slight superior and lateral angle.
  Patients will be educated on how to perform the 7 sets of frozen shoulder exercise. Subjects will be advised to perform all the exercises to a point that they may feel tightness but not painful and hold to the point for 2-3 seconds.
Device: App-assisted exercise — Patients will be educated on how to perform the 7 sets of frozen shoulder exercise. Subjects will be advised to perform all the exercises to a point that they may feel tightness but not painful and hold to the point for 2-3 seconds. Then the APP group will suggest performing the exercise from APP education The APP intervention group will be guided through the exercises using the mobile app, while the conventional group will be provided with a printed pamphlet illustrating the exercises.. Each set exercise will have 10 repetitions and investigators recommend 4 sessions per day.
  Arms: App intervention group
Drug: Nonsteroidal anti-inflammatory drugs (aceclofenac) — All patients will be prescribed two weeks of nonsteroidal anti-inflammatory drugs (aceclofenac) .

SUMMARY:
Abstract

Introduction Frozen shoulder is a common musculoskeletal disorder with reported lifetime prevalence to be 2%~5% in the general population. Patients with frozen shoulders present with chronic pain and limited range of motion of affected shoulder and often cause an adverse impact on their daily activities and working ability. Shoulder exercises had been proven to be effective in treatment of frozen shoulders and the effects were even better after intraarticular corticosteroid injection. Strategies to enhance home exercise for patients with frozen shoulders are essential.

Objective To compare the effects of home exercises delivered by a newly developed app named Defrozen app with that by convention home exercise for frozen shoulder patients after intra-articular corticosteroid injection.

Methods and analysis This is a randomized, controlled, assessor-blinded clinical trial. Seventy-eight individuals diagnosed with frozen shoulders will be randomly divided into two groups. The primary outcome will be shoulder passive range of motion (measured with a universal goniometer). The secondary outcomes will include , shoulder pain evaluated by 11-point numeric rating scale , Oxford shoulder score and Disabilities of the arm, shoulder and hand questionnaire. Feasibility of the app includes including Technology Acceptance Model (TAM-2), System Usability Scale (SUS) and Usability, Satisfaction and Ease of Use (USE) questionnaire . The treatment will be conducted for 6 months (Defrozen app home exercise x conventional home exercise by instructions from printed pamphlets).All participants will receive outcome measurements assessment prior to randomization , 4 weeks , 12 weeks after injections interventions. Feasibility will be evaluated 4 weeks after intervention in the Defrozen app group.

Ethics and dissemination The study protocol was approved by the Institutional Review Board. The findings of the trial will be disseminated through peer-reviewed journals and scientific conferences.

DETAILED DESCRIPTION:
The primary objective of this study is to test the hypothesis that a 12-week frozen shoulder exercise program delivered through the mobile app will result in greater improvement in shoulder range of motion compared to the control group. The control group will receive conventional home exercises provided on paper for patients with frozen shoulder after undergoing intra-articular corticosteroid injection.The secondary objective is to assess the differences in range of motion and functional outcomes between the two groups of patients. Additionally, the feasibility and acceptability of the Defrozen-App to these patients will be evaluated.

This study will employ a prospective, two-armed, assessor-blinded superiority randomized controlled trial design to compare two parallel groups of patients with primary frozen shoulder. The study was designed in accordance with the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) guidelines for planning interventional trials. The trial results will be reported following the Consolidated Standards of Reporting Trials (CONSORT) guidelines.

This study will be conducted in the northern branch of a medical system, which includes three hospitals located in northern Taiwan. The trial is registered [provide registration number or leave it blank if not available]. The recruitment of patients will take place in the clinic of the Department of Physical Medicine and Rehabilitation at Chang Gung Memorial Hospital, Taipei, Linko, and Taoyuan branches.

A Mobile Phone App for Demonstrating Home Exercises for Frozen Shoulder:

The Defrozen app is designed to provide simple home exercise programs for patients with frozen shoulders. It includes various features such as a training mode with exercise demonstrations, an exercise calendar, and pain evaluation.The main screen of the app displays exercise videos that are demonstrated by one of our researchers. It consists of seven sets of exercises specifically selected by physicians and a physiotherapist in our team. These exercises include Finger Walk for shoulder flexion and abduction, self-stretching exercises for shoulder external rotation and pectoral muscles, and crossover arm stretch for shoulder adduction. Additionally, towel exercises for shoulder extension and internal rotation are included. Each set of exercises consists of 10 repetitions, and we recommend performing four sessions per day. The total exercise time for one session is approximately 8 minutes. We encourage users to follow the exercise demonstrations provided in the app.After completing the exercise mode, the app prompts the patient to indicate whether they have completed the exercise and record their current pain intensity on a scale ranging from 0 to 10 . The app then transitions to the calendar mode, which displays the number of exercise sessions completed on that day and reminds the patient of the remaining sessions to be completed.

Procedures:

Participants will be recruited from the clinics of physical medicine and rehabilitation in a medical center located in northern Taiwan. Detailed information about the study will be provided to all eligible patients, and written informed consent will be obtained from each participant. All study visits will take place at a clinical laboratory near the clinics.

The assessor will collect baseline data from participants prior to randomization. Follow-up assessments will be conducted at two time points: 4 weeks after the interventions and 12 weeks after the interventions. Feasibility of the interventions will be evaluated only after the 4-week intervention period.

Random Allocation:

Random allocation of participants will be conducted using computer-generated random numbers in a 1:1 ratio. This process will be performed by one of the authors who is independent of the screening, patient recruitment, clinical care, and data collection. Subjects will be randomly assigned to either the Defrozen App group or the conventional group, ensuring equal allocation between the two groups.

The generated random number list will be placed into sequentially numbered, opaque, and sealed envelopes. These envelopes will be securely stored by the researcher responsible for allocation. Once a subject has been confirmed as eligible and has provided informed consent, the envelope corresponding to their sequential order will be opened to reveal their group allocation.

Blinding:

Participant allocation and follow-up arrangements will be overseen by a clinical researcher who will not be blinded to the participants' group assignments. However, to minimize bias, outcome measure assessments will be conducted by a physician from the study team who will be unaware of the participants' intervention groups.

Interventions In this study, all patients, regardless of their group allocation, will receive both glenohumeral joint and subacromial space injections. This decision is based on previous research that has suggested a synergistic effect of combination injections in increasing joint internal rotation angle. (Proper site of corticosteroid injection for the treatment of idiopathic frozen shoulder: Results from a randomized trial)The injections will consist of a solution containing 1 ml of 40 mg/ml triamcinolone acetonide and 1 ml of 1% lidocaine in each site. The glenohumeral joint injection will be performed blindly using an anterior approach. The needle will be inserted medially to the head of the humerus, located approximately 1 cm lateral to the coracoid process, and directed posteriorly at a slight superior and lateral angle.Previous studies have suggested that blind anterior glenohumeral joint injection yields comparable pain and functional outcomes to ultrasound-guided injection. Additionally, the anterior approach has shown better pain control and improved functional activity recovery in the early stages of primary frozen shoulder compared to the posterior approach.

For the subacromial injection, ultrasound guidance will be employed to potentially achieve greater clinical improvement in shoulder pain compared to blind injection.Following the injections, patients will receive instructions on performing the seven sets of frozen shoulder exercises mentioned earlier. The APP group will be guided through the exercises using the mobile app, while the conventional group will be provided with a printed pamphlet illustrating the exercises. Each set of exercises will involve 10 repetitions, and it is recommended to perform four sessions per day. Additionally, all patients will be prescribed two weeks of nonsteroidal anti-inflammatory drugs (aceclofenac) to manage pain and inflammation.

ELIGIBILITY:
Eligibility Criteria:

Patients with frozen shoulder who are scheduled to receive intra-articular glucocorticosteroid injections, as determined by the physician investigator, will be consecutively enrolled in the study. To be included in the study, patients must meet the following criteria:

1. Unilateral frozen shoulder.
2. Suitability for treatment with intra-articular and subacromial glucocorticosteroid injection.
3. Patients must fulfill the diagnostic criteria for frozen shoulder, as described by Bulgen et al. These criteria include shoulder pain persisting for at least 1 month, sleep disturbance (such as night pain or inability to lie on the affected side), restriction of all active and passive shoulder movements, and a reduction of passive glenohumeral external rotation by at least 50% compared to the unaffected side.
4. Plain radiographs of the shoulder will be obtained to exclude other pathologies.

Patients will be excluded from the study if they meet any of the following criteria:

1. Age younger than 20 years old.
2. Bilateral involvement of the shoulder.
3. Secondary frozen shoulder resulting from trauma.
4. History of shoulder joint injections or upper limb surgery within the past month.

   Presence of rheumatoid arthritis, central nervous system disorders, or cervical radiculopathy.
5. Cognitive disorders or inability to understand exercise instructions.
6. Contraindications for anesthesia or corticosteroid injection.
7. Lack of familiarity with using smartphones.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-09-11 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change shoulder active range of motion in degree | prior to randomization, 4-weeks after interventions and 12-weeks after intervention
  The range of motion of the shoulder will be assessed using a universal goniometer, which measures the angle of movement between specific bone landmarks. The investigator will evaluate the active range of motion of the affected shoulder, including flexion, abduction, internal rotation, and external rotation, using the goniometer to determine the degrees of movement in each direction. Active range of movement of the affected shoulder, including flexion, abduction, internal rotation, and external rotation, will be measured by goniometer in degree.

SECONDARY OUTCOMES:
Change of Shoulder pain by Numeric Rating Scale (NRS) | prior to randomization, 4-weeks after interventions and 12-weeks after intervention
  To assess shoulder pain, investigators will utilize an 11-point NRS. Patients will be informed that a score of 0 represents no pain, while a score of 10 indicates the highest level of pain.
Change of Oxford shoulder score (OSS). | prior to randomization, 4-weeks after interventions and 12-weeks after intervention
  A patient-rated outcome measure of shoulder pain and function in patients with shoulder pain. OSS has twelve questions with five possible responses ranging from 0 (worst) to 4 (best).
Change of Quick Disability of the Arm, Shoulder and Head (QuickDASH) score | prior to randomization, 4-weeks after interventions and 12-weeks after intervention
  The QuickDASH is a modified version of the original 30-item Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire, consisting of 11 items. A minimum of 10 items must be completed by the participant. Each item has five response options.The total QuickDASH score ranges from 0 (indicating no disability) to 100 (representing the most severe disability)
Selected part of revised Technology Acceptance Model (TAM-2) | 4 weeks after intervention in App intervention group
  The selected part of revised Technology Acceptance Model(TAM-2) including intention to use, perceived usefulness and perceived ease of use. Participants will be asked to rate their agreement with each statement on a five-point Likert scale, ranging from "Strongly Disagree" to "Strongly Agree."
System Usability Scale (SUS) | 4 weeks after intervention in App intervention group
  he SUS is a standardized questionnaire that consists of ten statements related to the usability of the application. Participants will be asked to rate their agreement with each statement on a five-point Likert scale, ranging from "Strongly Disagree" to "Strongly Agree."
Usability, Satisfaction and Ease of Use (USE) questionnaire | 4 weeks after intervention in App intervention group
  The questionnaire consists of four statements related to the system or application being evaluated. Participants will be asked to rate their agreement with each statement on a five-point Likert scale, ranging from "Strongly Disagree" to "Strongly Agree."

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chi Chen, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mezian K, Coffey R, Chang KV. Frozen Shoulder(Archived). 2023 Aug 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482162/ PMID 29489251
- [Background] Walker-Bone K, Palmer KT, Reading I, Coggon D, Cooper C. Prevalence and impact of musculoskeletal disorders of the upper limb in the general population. Arthritis Rheum. 2004 Aug 15;51(4):642-51. doi: 10.1002/art.20535. PMID 15334439
- [Background] Sarasua SM, Floyd S, Bridges WC, Pill SG. The epidemiology and etiology of adhesive capsulitis in the U.S. Medicare population. BMC Musculoskelet Disord. 2021 Sep 27;22(1):828. doi: 10.1186/s12891-021-04704-9. PMID 34579697
- [Background] Millar NL, Meakins A, Struyf F, Willmore E, Campbell AL, Kirwan PD, Akbar M, Moore L, Ronquillo JC, Murrell GAC, Rodeo SA. Frozen shoulder. Nat Rev Dis Primers. 2022 Sep 8;8(1):59. doi: 10.1038/s41572-022-00386-2. PMID 36075904
- [Background] Mertens MG, Meert L, Struyf F, Schwank A, Meeus M. Exercise Therapy Is Effective for Improvement in Range of Motion, Function, and Pain in Patients With Frozen Shoulder: A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2022 May;103(5):998-1012.e14. doi: 10.1016/j.apmr.2021.07.806. Epub 2021 Aug 21. PMID 34425089
- [Background] Russell S, Jariwala A, Conlon R, Selfe J, Richards J, Walton M. A blinded, randomized, controlled trial assessing conservative management strategies for frozen shoulder. J Shoulder Elbow Surg. 2014 Apr;23(4):500-7. doi: 10.1016/j.jse.2013.12.026. PMID 24630545
- [Background] Robinson PM, Norris J, Roberts CP. Randomized controlled trial of supervised physiotherapy versus a home exercise program after hydrodilatation for the management of primary frozen shoulder. J Shoulder Elbow Surg. 2017 May;26(5):757-765. doi: 10.1016/j.jse.2017.01.012. Epub 2017 Mar 18. PMID 28318848
- [Background] Challoumas D, Biddle M, McLean M, Millar NL. Comparison of Treatments for Frozen Shoulder: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Dec 1;3(12):e2029581. doi: 10.1001/jamanetworkopen.2020.29581. PMID 33326025
- [Background] Pandey V, Madi S. Clinical Guidelines in the Management of Frozen Shoulder: An Update! Indian J Orthop. 2021 Feb 1;55(2):299-309. doi: 10.1007/s43465-021-00351-3. eCollection 2021 Apr. PMID 33912325
- [Background] Gleyze P, Clavert P, Flurin PH, Laprelle E, Katz D, Toussaint B, Benkalfate T, Charousset C, Joudet T, Georges T, Hubert L, Lafosse L, Hardy P, Solignac N, Levigne C; French Arthroscopy Society. Management of the stiff shoulder. A prospective multicenter comparative study of the six main techniques in use: 235 cases. Orthop Traumatol Surg Res. 2011 Dec;97(8 Suppl):S167-81. doi: 10.1016/j.otsr.2011.09.004. Epub 2011 Oct 28. PMID 22036993
- [Background] Hardage J, Peel C, Morris D, Graham C, Brown C, Foushee HR, Braswell J. Adherence to Exercise Scale for Older Patients (AESOP): a measure for predicting exercise adherence in older adults after discharge from home health physical therapy. J Geriatr Phys Ther. 2007;30(2):69-78. doi: 10.1519/00139143-200708000-00006. PMID 18171490
- [Background] Chen HC, Chuang TY, Lin PC, Lin YK, Chuang YH. Effects of Messages Delivered by Mobile Phone on Increasing Compliance With Shoulder Exercises Among Patients With a Frozen Shoulder. J Nurs Scholarsh. 2017 Jul;49(4):429-437. doi: 10.1111/jnu.12308. Epub 2017 Jun 20. PMID 28632975
- [Background] Liao CH, Wu YT, Cheng CT, Ooyang CH, Kang SC, Fu CY, Hsu YP, Hsieh CH, Chen CC. An Image-Based Mobile Health App for Postdrainage Monitoring: Usability Study. J Med Internet Res. 2020 Aug 28;22(8):e17686. doi: 10.2196/17686. PMID 32857060
- [Background] Pfeifer AC, Uddin R, Schroder-Pfeifer P, Holl F, Swoboda W, Schiltenwolf M. Mobile Application-Based Interventions for Chronic Pain Patients: A Systematic Review and Meta-Analysis of Effectiveness. J Clin Med. 2020 Nov 5;9(11):3557. doi: 10.3390/jcm9113557. PMID 33167300
- [Background] Steiner B, Richter I, Elgert L, Haux R, Wolf KH. Mobile Health Applications for Rehabilitation of Musculoskeletal Diseases of the Shoulder: A Systematic Analysis. Stud Health Technol Inform. 2021 May 24;278:195-202. doi: 10.3233/SHTI210069. PMID 34042894
- [Background] Elgert L, Steiner B, Saalfeld B, Marschollek M, Wolf KH. Health-Enabling Technologies to Assist Patients With Musculoskeletal Shoulder Disorders When Exercising at Home: Scoping Review. JMIR Rehabil Assist Technol. 2021 Feb 4;8(1):e21107. doi: 10.2196/21107. PMID 33538701
- [Background] Carbonaro N, Lucchesi I, Lorusssi F, Tognetti A. Tele-monitoring and tele-rehabilitation of the shoulder muscular-skeletal diseases through wearable systems. Annu Int Conf IEEE Eng Med Biol Soc. 2018 Jul;2018:4410-4413. doi: 10.1109/EMBC.2018.8513371. PMID 30441330
- [Background] Stutz T, Emsenhuber G, Huber D, Domhardt M, Tiefengrabner M, Oostingh GJ, Fotschl U, Matis N, Ginzinger S. Mobile Phone-Supported Physiotherapy for Frozen Shoulder: Feasibility Assessment Based on a Usability Study. JMIR Rehabil Assist Technol. 2017 Jul 20;4(2):e6. doi: 10.2196/rehab.7085. PMID 28729234
- [Background] Choi Y, Nam J, Yang D, Jung W, Lee HR, Kim SH. Effect of smartphone application-supported self-rehabilitation for frozen shoulder: a prospective randomized control study. Clin Rehabil. 2019 Apr;33(4):653-660. doi: 10.1177/0269215518818866. Epub 2018 Dec 10. PMID 30526016
- [Background] Bulgen DY, Binder AI, Hazleman BL, Dutton J, Roberts S. Frozen shoulder: prospective clinical study with an evaluation of three treatment regimens. Ann Rheum Dis. 1984 Jun;43(3):353-60. doi: 10.1136/ard.43.3.353. PMID 6742895
- [Background] Kelley MJ, Shaffer MA, Kuhn JE, Michener LA, Seitz AL, Uhl TL, Godges JJ, McClure PW. Shoulder pain and mobility deficits: adhesive capsulitis. J Orthop Sports Phys Ther. 2013 May;43(5):A1-31. doi: 10.2519/jospt.2013.0302. Epub 2013 Apr 30. No abstract available. PMID 23636125
- [Background] Mintken PE, Glynn P, Cleland JA. Psychometric properties of the shortened disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH) and Numeric Pain Rating Scale in patients with shoulder pain. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):920-6. doi: 10.1016/j.jse.2008.12.015. Epub 2009 Mar 17. PMID 19297202
- [Background] Dawson J, Fitzpatrick R, Carr A. Questionnaire on the perceptions of patients about shoulder surgery. J Bone Joint Surg Br. 1996 Jul;78(4):593-600. PMID 8682827
- [Background] Dawson J, Rogers K, Fitzpatrick R, Carr A. The Oxford shoulder score revisited. Arch Orthop Trauma Surg. 2009 Jan;129(1):119-23. doi: 10.1007/s00402-007-0549-7. Epub 2008 Jan 9. PMID 18183410
- [Background] Rangan A, Brealey SD, Keding A, Corbacho B, Northgraves M, Kottam L, Goodchild L, Srikesavan C, Rex S, Charalambous CP, Hanchard N, Armstrong A, Brooksbank A, Carr A, Cooper C, Dias JJ, Donnelly I, Hewitt C, Lamb SE, McDaid C, Richardson G, Rodgers S, Sharp E, Spencer S, Torgerson D, Toye F; UK FROST Study Group. Management of adults with primary frozen shoulder in secondary care (UK FROST): a multicentre, pragmatic, three-arm, superiority randomised clinical trial. Lancet. 2020 Oct 3;396(10256):977-989. doi: 10.1016/S0140-6736(20)31965-6. PMID 33010843
- [Background] Sharma SP, Baerheim A, Kvale A. Passive range of motion in patients with adhesive shoulder capsulitis, an intertester reliability study over eight weeks. BMC Musculoskelet Disord. 2015 Feb 22;16:37. doi: 10.1186/s12891-015-0495-4. PMID 25888419
- [Background] Beaton DE, Wright JG, Katz JN; Upper Extremity Collaborative Group. Development of the QuickDASH: comparison of three item-reduction approaches. J Bone Joint Surg Am. 2005 May;87(5):1038-46. doi: 10.2106/JBJS.D.02060. PMID 15866967
- [Background] Gummesson C, Ward MM, Atroshi I. The shortened disabilities of the arm, shoulder and hand questionnaire (QuickDASH): validity and reliability based on responses within the full-length DASH. BMC Musculoskelet Disord. 2006 May 18;7:44. doi: 10.1186/1471-2474-7-44. PMID 16709254
- [Background] Liang HW, Wang HK, Yao G, Horng YS, Hou SM. Psychometric evaluation of the Taiwan version of the Disability of the Arm, Shoulder, and Hand (DASH) questionnaire. J Formos Med Assoc. 2004 Oct;103(10):773-9. PMID 15490028
- [Background] Vorrink SN, Kort HS, Troosters T, Lammers JW. A Mobile Phone App to Stimulate Daily Physical Activity in Patients with Chronic Obstructive Pulmonary Disease: Development, Feasibility, and Pilot Studies. JMIR Mhealth Uhealth. 2016 Jan 26;4(1):e11. doi: 10.2196/mhealth.4741. PMID 26813682
- [Background] Cho CH, Kim du H, Bae KC, Lee D, Kim K. Proper site of corticosteroid injection for the treatment of idiopathic frozen shoulder: Results from a randomized trial. Joint Bone Spine. 2016 May;83(3):324-9. doi: 10.1016/j.jbspin.2015.06.014. Epub 2016 Feb 10. PMID 26875065
- [Background] Tallia AF, Cardone DA. Diagnostic and therapeutic injection of the shoulder region. Am Fam Physician. 2003 Mar 15;67(6):1271-8. PMID 12674455
- [Background] Cho CH, Min BW, Bae KC, Lee KJ, Kim DH. A prospective double-blind randomized trial on ultrasound-guided versus blind intra-articular corticosteroid injections for primary frozen shoulder. Bone Joint J. 2021 Feb;103-B(2):353-359. doi: 10.1302/0301-620X.103B2.BJJ-2020-0755.R1. PMID 33517741
- [Background] Deng Z, Li Z, Li X, Chen Z, Shen C, Sun X, Shu H, Wu J, Tang K. Comparison of Outcomes of Two Different Corticosteroid Injection Approaches for Primary Frozen Shoulder: A Randomized Controlled Study. J Rehabil Med. 2023 Jan 3;55:jrm00361. doi: 10.2340/jrm.v55.2201. PMID 36597664
- [Background] Wu T, Song HX, Dong Y, Li JH. Ultrasound-guided versus blind subacromial-subdeltoid bursa injection in adults with shoulder pain: A systematic review and meta-analysis. Semin Arthritis Rheum. 2015 Dec;45(3):374-8. doi: 10.1016/j.semarthrit.2015.05.011. Epub 2015 May 21. PMID 26590864
- [Background] Antoine Parker C, Ellis R. Effect of Electronic Messaging on Physical Activity Participation among Older Adults. J Aging Res. 2016;2016:6171028. doi: 10.1155/2016/6171028. Epub 2016 May 17. PMID 27293891
- [Background] Kim BH, Glanz K. Text messaging to motivate walking in older African Americans: a randomized controlled trial. Am J Prev Med. 2013 Jan;44(1):71-5. doi: 10.1016/j.amepre.2012.09.050. PMID 23253653